CLINICAL TRIAL: NCT00071461
Title: A Double-blind, Randomized, Placebo-controlled, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of Bosentan in Patients With Idiopathic Pulmonary Fibrosis, Open Label Extension
Brief Title: Efficacy and Safety of Oral Bosentan in Patients With Idiopathic Pulmonary Fibrosis
Acronym: BUILD 1
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-320; BUILD 1
Record Dates: First submitted 2003-10-23; First posted 2003-10-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; Interstitial lung disease; Bosentan; BUILD
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Initial dose: 62.5 mg b.i.d. for 4 weeks.
  * Target dose: - body weight > 40 kg (90 lb): 125 mg b.i.d., (if the initial dose is well tolerated).
  * body weight < 40 kg (90 lb): 62.5 mg b.i.d.
  Interventions: Drug: bosentan
- 2 (Placebo Comparator): Initial dose: 62.5 mg b.i.d. for 4 weeks.
  * Target dose: - body weight > 40 kg (90 lb): 125 mg b.i.d., (if the initial dose is well tolerated).
  * body weight < 40 kg (90 lb): 62.5 mg b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bosentan — Initial dose: 62.5 mg b.i.d. for 4 weeks.
  * Target dose: - body weight > 40 kg (90 lb): 125 mg b.i.d., (if the initial dose is well tolerated).
  * body weight < 40 kg (90 lb): 62.5 mg b.i.d.
  Other Names: Tracleer
  Arms: 1
Drug: Placebo — Initial dose: 62.5 mg b.i.d. for 4 weeks.
  * Target dose: - body weight > 40 kg (90 lb): 125 mg b.i.d., (if the initial dose is well tolerated).
  * body weight < 40 kg (90 lb): 62.5 mg b.i.d.
  Arms: 2

SUMMARY:
Endothelin-1 (ET-1) is expressed in a variety of pulmonary pathological conditions including pulmonary vascular disease and pulmonary fibrosis.

Bosentan (an oral dual ET-1 receptor antagonist) could delay the progression of idiopathic pulmonary fibrosis (IPF), a condition for which no established treatment is available.

The present trial investigates a possible use of bosentan, which is currently approved for the treatment of symptoms of pulmonary arterial hypertension (PAH) WHO class III and IV, to a new category of patients suffering from IPF.

It was decided to offer Open Label treatment (bosentan) for patients willing to continue in the BUILD 1 study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 18 years of age.

   * Women must be either postmenopausal (i.e., amenorrhea for at least 1 year), or surgically or naturally sterile.
   * Women of childbearing potential must have a negative pre-treatment pregnancy test and use a reliable method of contraception during study treatment and for at least 3 months after study treatment termination.
2. IPF proven diagnosis < 3 years documented according to ATS/ERS international multidisciplinary consensus, with or without surgical (thoracoscopic or open) chest lung biopsy
3. Duration of illness ≥ 3 months.
4. Six-minute walk test distance (limited by dyspnea) ≥ 150 meters and < 500 meters
5. Patients who have signed the informed consent form prior to initiation of any study procedure.

Exclusion Criteria:

1. Interstitial lung disease due to conditions other than IPF, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans with organizing pneumonia, and cancer.
2. History of clinically significant environmental exposure known to cause pulmonary fibrosis (drugs, asbestos, beryllium, radiation, domestic birds, etc.).
3. Severe concomitant illness limiting life expectancy (< 1 year).
4. FVC ≥ 90% predicted.
5. Severe restrictive lung disease: FVC < 50% predicted or FVC < 1.2 l, or DLco < 30% predicted or residual volume ≥ 120% predicted.
6. Severe obstructive lung disease: FEV1/FVC< 0.65.
7. Documented improvement of patient's condition within 12 months prior to randomization with or without IPF-specific therapy (e.g., corticosteroids, immunosuppressive, cytotoxic or antifibrotic drugs, TNFa blocker, interferon g).
8. Recent pulmonary or upper respiratory track infection (within 4 weeks of randomization).
9. PaO2 < 55 mm Hg (sea level) or 50 mm Hg (altitude) at rest on room air.
10. Echocardiographic evidence of severe pulmonary hypertension (PH): systolic pulmonary pressure ≥ 50 mm Hg or tricuspid regurgitation velocity ≥ 3.2 m/sec (unless severe PH is invalidated by a right heart catheterization). If the pulmonary pressure is not quantifiable, presence of significant right ventricular enlargement or hypertrophy or right ventricular dysfunction.
11. Severe chronic heart failure, e.g., NYHA class III or IV and/or left ventricular ejection fraction < 25%.
12. Acute or chronic impairment (other than dyspnea) limiting the ability to comply with study requirements, e.g., the 6MWT or the PFTs.

    (e.g., angina pectoris, intermittent claudicating, chronic arthritis).
13. Baseline values of liver transaminases, i.e., aspartate aminotransferases (AST) and/or alanine aminotransferases (ALT) > 3 times the upper limit of normal ranges.
14. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C.
15. Serum creatinine ≥ 2.5 mg/dl (221 mmol/l) or dialysis.
16. Hemoglobin concentration < 75% the lower limit of normal ranges.
17. Systolic blood pressure < 85 mm Hg.
18. Pregnancy or breast-feeding.
19. Current drug or alcohol dependence.
20. Smoker (≥ 5 cigarettes per day) or former smoker (≥ 5 cigarettes per day) having stopped less than 6 months prior to randomization.
21. Recently started (< 8 weeks from Screening visit) or planned cardio-pulmonary rehabilitation program based on exercise.
22. Treatment with oral corticosteroids (> 15 mg/day prednisone or equivalent), immunosuppressive, cytotoxic or antifibrotic drugs such as TNF alpha blocker, or interferon gamma within 4 weeks of randomization.within 4 weeks of randomization.
23. Treatment with glibenclamide (glyburide), cyclosporine A or tacrolimus within 1 weeks of randomization.
24. Treatment with an endothelin receptor antagonist within 3 months of randomization.
25. Treatment within 3 months of randomization or planned treatment with another investigational drug.
26. Known hypersensitivity to bosentan or any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2003-08; Primary Completion 2005-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Change in 6-minute walk distance | Baseline to End-of-Period 1

SECONDARY OUTCOMES:
Death or treatment failure | Up to End-of-Period 1

CONTACTS AND LOCATIONS:
Locations (29):
- United States (16):
  - University of Alabama at Birmingham - Pulmonary Division, Birmingham, Alabama
  - David Geffen School of Medicine at UCLA - Division of Pulmonary and Critical Care Medicine, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - University of California - Ambulatory Care Center, San Francisco, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Jackson Memorial Hospital, Miami, Florida
  - University of Iowa Hospitals & Clinics - Department of Internal Medicine, Iowa City, Iowa
  - University of Michigan Health System - Division of Pulmonary & Critical Care Medicine, Ann Arbor, Michigan
  - Mayo Medical School - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Washington - Division of Pulmonary & Critical Care Medicine, Seattle, Washington
  - University of Wisconsin Hospitals & Clinics - Section of Pulmonary and Critical Care Medicine, Madison, Wisconsin
- Canada (3):
  - University of British Columbia - St. Paul's Hospital, Vancouver, British Columbia
  - Rosedale Medical Center, Toronto, Ontario
  - Notre-Dame Hospital - Clinique du Thorax, Montreal, Quebec
- France (3):
  - Hôpital Avicenne - Université de Paris, Bobigny
  - Médecine Spécialisée Aigüe - CHU Grenoble, Grenoble
  - Hôpital Louis Pradel, Lyon
- Germany (3):
  - Abt. Pneumologie Medizinische Klinik Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Klinik Löwenstein gGmbH, Löwenstein
  - Medizinische Klinik und Poliklinik I Klinikum der Universität München, München
- Sheba Medical Center, Tel Litwinsky, Israel
- Section of Respiratory Diseases - Policlinico Le Scotte - Siena University, Siena, Italy
- Inselspital, Bern, Switzerland
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Raghu G, King TE Jr, Behr J, Brown KK, du Bois RM, Leconte I, Roux S, Swigris J. Quality of life and dyspnoea in patients treated with bosentan for idiopathic pulmonary fibrosis (BUILD-1). Eur Respir J. 2010 Jan;35(1):118-23. doi: 10.1183/09031936.00188108. Epub 2009 Aug 13. PMID 19679600
- [Derived] King TE Jr, Behr J, Brown KK, du Bois RM, Lancaster L, de Andrade JA, Stahler G, Leconte I, Roux S, Raghu G. BUILD-1: a randomized placebo-controlled trial of bosentan in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2008 Jan 1;177(1):75-81. doi: 10.1164/rccm.200705-732OC. Epub 2007 Sep 27. PMID 17901413